CLINICAL TRIAL: NCT07219069
Title: Bispectral Monitoring on Mechanically Ventilated Patients, a Randomized Clinical Trial. (BIMV Trial)
Brief Title: Bispectral Monitoring on Mechanically Ventilated Patients
Acronym: BIMV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Pascal Kingah, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-25-0240
Record Dates: First submitted 2025-10-06; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Sedation
Keywords: sedation; Bispectral Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BIS group (Experimental)
  Interventions: Device: BIS group
- Non-BIS group (Active Comparator)
  Interventions: Other: Non-BIS group

INTERVENTIONS:
Device: BIS group — Participants will be placed on BIS monitoring continuously until extubation, transfer to another facility, change in status to comfort measures, or if the patient expires. The BIS monitoring system offers a continuous processed electroencephalographic measurement used to assess cerebral activity and can monitor the electrophysiologic effects of sedation and anesthetics.BIS monitoring offers numerical values which have been validated to reflect various sedation levels. BIS levels range from 0 to 100 with greater than 100 corresponding to wakefulness. Values less than 60 indicate deep sedation and values less than 40 correspond to deep anesthesia
  Arms: BIS group
Other: Non-BIS group — The usual protocol for titrating sedation will be followed using various sedation assessment scales such as Richmond Agitation Sedation Scale (RASS), Visual Analog Scale (VAS), Ramsay Sedation Scale (RSS), or Sedation Agitation Scale (SAS) per physicians choice.
  Arms: Non-BIS group

SUMMARY:
The purpose of this study is to determine the difference in the duration of mechanical ventilation, to evaluate the difference in ICU length of stay and to determine the difference in the overall dose of sedation medications between the between participants who were monitored using Bispectral index monitoring (BIS) monitors and those who were not.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the medical ICU
* Intubated on mechanical ventilation
* On sedation medication infusion

Exclusion Criteria:

* Patients with a history of chronic opioid use
* Patients with end-stage liver disease at ICU admission (i.e., International normalized ratio >1.5 and not taking warfarin and/or a total serum bilirubin 1.5 times above normal limits)
* Pregnant patients
* Current prisoner
* Refractory shock: Mean arterial blood pressure below 65 millimeters of mercury(65mmHg) despite maximum doses of 3 pressors. Norepinephrine 70mcg/min; vasopressin 0.03 units/min; epinephrine 35mcg/min; dopamine 20mcg/kg/min and phenylephrine 350mcg/min
* Inability to complete the required time for follow-up
* Surgical admission diagnosis
* Patients with skin conditions precluding BIS monitor sensor adherence
* Patients on neuromuscular blockade infusion or benzodiazepine infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Median ventilator time reported in hours | from the time the patient was intubated to the time they were extubated, changed to comfort measures, transferred to another facility, or expired(about 4-6 days)

SECONDARY OUTCOMES:
ICU length of stay | During ICU discharge or transfer out of ICU (about 5-7 days after admission to ICU)
Amount of sedation medication used | From start of ventilation to end of ventilation (about 4-6 days)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal L Kingah, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No